CLINICAL TRIAL: NCT02914860
Title: Comparison of the Ganglionated Plexi Activity in Patients With Different Forms of Atrial Fibrillation Guided by SUMO Technology
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Spectrum Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Volunteers+AF patients
Record Dates: First submitted 2016-09-08; First posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Volunteers (Experimental): Healthy volunteers
  Interventions: Device: Cardiac CT; Device: D-SPECT
- PAF (Active Comparator): Patients with paroxysmal atrial fibrillation
  Interventions: Device: Cardiac CT; Procedure: Ablation Procedure; Device: D-SPECT
- Pers AF (Active Comparator): Patients with persistent atrial fibrillation
  Interventions: Device: Cardiac CT; Procedure: Ablation Procedure; Device: D-SPECT
- L-s Pers AF (Active Comparator): Patients with long-standing persistent atrial fibrillation
  Interventions: Device: Cardiac CT; Procedure: Ablation Procedure; Device: D-SPECT

INTERVENTIONS:
Device: Cardiac CT — * Cardiac CT - contract enhanced cardiac CT according to standard protocol
  * D-SPECT SUMO study - standard SUMO protocol (suggested reduction in mIBG dose and increase in scan time to minimize overall radiation burden)
  * Merge CT and D-SPECT image data to generate SUMO map.
Procedure: Ablation Procedure — 1. CARTO-reconstruction LA, preferably during same rhythm as SUMO map (generally sinus rhythm) for use during registration of SUMO map in CARTO.
  2. High frequency stimulation (HFS; 20-Hz frequency, 5-ms pulse duration, and 15-mA output) to access positive vagal response (the heart rate decreasing by 50% at baseline).
  3. RF ablation only at points where there is an HFS positive response to SUMO DUA (in sinus rhythm if AF converts)
  4. Target a region of 1.0 - 1.5 cm diameter around the SUMO mIBG DUA
  5. Control HFS
  6. At operator discretion, conventional PVI by circumferential antral ablation according to standard procedures.
  7. Exit and entrance block confirmation
  8. Attempt to induce sustained atrial tachycardia; optional mapping and ablation of post-ablation atrial tachycardia.
  Arms: L-s Pers AF; PAF; Pers AF
Device: D-SPECT

SUMMARY:
The purpose of this study is to compare DUA (discrete uptake accumulations) of mIBG activity in patients with different forms of atrial fibrillation and within a sub-group of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age ≥ 18 and ≤ 80 years.
2. Male or female, age ≥ 50 years in the healthy volunteers group
3. No heart pathology (for volunteers)
4. PAF, Pers AF and L-s Pers AF (ECG documented).
5. LVEF ≥ 50%
6. Able to provide written informed consent
7. Able to comply with the requirements of the study

Exclusion Criteria:

1. Previous AF ablation therapy
2. Clinical evidence of active coronary ischemia, significant valvular heart disease, or hemodynamically significant congenital cardiac abnormality
3. Recent (3 months) myocardial infarction (MI), stroke or transient ischemic attack (except if the patient had a DES implanted stent post-MI it would be one year)
4. Contra-indication to Iodine-123 Meta-iodobenzylguanidine (123I-mIBG), iodine, isoproterenol
5. Use of medication for non-cardiac medical conditions that is known to interfere with 123I-mIBG uptake and cannot be safely withheld for at least 24 hours prior to the D-SPECT study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
location of discrete uptake accumulations | 1 week

SECONDARY OUTCOMES:
adverse events | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia